CLINICAL TRIAL: NCT05409885
Title: Comparison of the Effect of General and Spinal Anesthesia on Umbilical Neutrophil-to-lymphocyte Ratio, Platelet-to-lymphocyte Ratio and Mean Platelet Volume in Patients Undergoing Cesarean Section
Brief Title: The Effect of General and Spinal Anesthesia on Neutrophil-to-lymphocyte Ratio
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 5/4
Record Dates: First submitted 2022-04-20; First posted 2022-06-08 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia, General; Anesthesia, Spinal; Umbilical Cord
Keywords: anesthesia; cesarean section; neutrophil-to-lymphocyte ratio; platelet-to-lymphocyte ratio; mean platelet volume
MeSH Terms: interventions — Anesthesia, General; Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General anesthesia group: Evaluate the effects of general anesthesia on NLR, PLR and MPV in patients undergoing cesarean section.
  Interventions: Other: General anesthesia
- Spinal anesthesia group: Evaluate the effects of spinal anesthesia on NLR, PLR and MPV in patients undergoing cesarean section.
  Interventions: Other: Spinal anesthesia

INTERVENTIONS:
Other: General anesthesia — Evaluate the effects of general anesthesia on NLR, PLR and MPV in patients undergoing cesarean section.
  Groups: General anesthesia group
Other: Spinal anesthesia — Evaluate the effects of spinal anesthesia on NLR, PLR and MPV in patients undergoing cesarean section.
  Groups: Spinal anesthesia group

SUMMARY:
The aim of the study was to evaluate the effects of anesthetic techniques (general and spinal anesthesia) on umbilical cord neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR) and mean platelet volume (MPV) in patients undergoing cesarean section.

DETAILED DESCRIPTION:
This study was designed to evaluate the effects of anesthetic techniques (general and spinal anesthesia) on umbilical cord NLR, PLR and MPV in patients undergoing cesarean section.

The primary endpoint was to compare the effects of general and spinal anesthesia on umbilical cord NLR. Secondary endpoints were determined the general and spinal anesthesia on routine umbilical cord PLR, MPV and newborn Apgar scores at 1st and 5th min.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 45 years
* American Society of Anesthesiology (ASA) II-III
* elective ceserean surgery

Exclusion Criteria:

* declining to give written informed consent
* under 18 years of age or over 45 years of age
* factors affecting NLR, PLR and MPV such as preeclampsia, HELLP syndrome or premature rupture of membranes
* history of neurological and/or neuromucular disease
* cooperation cannot be established
* emergency surgery

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: elective ceserean surgery
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
neutrophil-to-lymphocyte ratio | within 5 minute, following delivery
  Evaluate the effects of NLR in patients undergoing cesarean section

SECONDARY OUTCOMES:
platelet-to-lymphocyte ratio | within 5 minute, following delivery
  Evaluate the effects of PLR in patients undergoing cesarean section
mean platelet volume | within 5 minute, following delivery
  Evaluate the effects of MPV in patients undergoing cesarean section
Newborn Apgar score 1st minute | 1st minute after birth
  Appearance (skin color), Pulse (heart rate), Grimace (reflex irritability), Activity (tone), Respiration. Apgar score at 1st min (0-3: severely depressed, 4-6: moderately depressed, 7-10: excellent condition)
Newborn Apgar score 5th minute | 5th minute after birth
  Appearance (skin color), Pulse (heart rate), Grimace (reflex irritability), Activity (tone), Respiration. Apgar score at 1st min (0-3: severely depressed, 4-6: moderately depressed, 7-10: excellent condition)

CONTACTS AND LOCATIONS:
Overall Officials: Kerem İnanoğlu, Principal Investigator — Antalya TRH; Esra Bağ, Principal Investigator — Antalya TRH; Arzu Karaveli, Study Director — Antalya TRH
Locations (1):
- Antalya Training and Research Hospital, Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No